CLINICAL TRIAL: NCT02774785
Title: Reducing Re-excisions After Breast Conserving Surgery: A Randomized Controlled Trial Comparing the MarginProbe Device in Addition to Standard Operating Procedure Versus Standard Operating Procedure Alone in Preventing Re-excision
Brief Title: Does Intra-operative MarginProbe Use Reduce Re-excision Rates?
Acronym: MarginProbe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 161393; PB-PG-0712-28108 (Other Grant/Funding Number: RfPB); 15-NW-0306 (Other: Research Ethics Committee)
Record Dates: First submitted 2016-03-22; First posted 2016-05-17 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device Arm (Experimental): Randomized for MarginProbe device to be used during surgical procedure
  Interventions: Device: MarginProbe
- Control Arm (No Intervention): Randomized for surgical procedure to happen as per standard care

INTERVENTIONS:
Device: MarginProbe — Surgery to take place as per standard care. When the surgery is nearly concluded, patient to be randomised. If randomised to device arm, the MarginProbe device will be used on the outer edge of the tumour and shavings. If the MarginProbe device indicates that cancer is detected, a further shaving is to be taken. Surgery then to be concluded as per standard care.
  Arms: Device Arm

SUMMARY:
The new device we are looking at is called the MarginProbe. It is a disposable probe which measures the margins of tissue removed to check they are clear of cancer cells, during breast conservation surgery. After specimen radiology, allows the Surgeon to remove further tissue if necessary, during the same operation if any involved margins are identified. This minimises the need for further repeat operations.

Previous studies carried out elsewhere in the world (USA and Israel) have identified that the probe reduces re-excision rate but there has never been a study in the UK.

The trial involves randomly allocating patients once they are in theatre, to either the MarginProbe procedure after breast conserving surgery and radiology has been completed, or not.

DETAILED DESCRIPTION:
Almost 60% of all patients diagnosed with breast cancer (48000 annually in the UK) undergo breast conserving surgery (BCS. Surgical removal of the cancer aims to reduce the risk of local recurrence and patient mortality. In order to minimise the amount of tissue removed, excision up to the cancer-free area (margins) is undertaken. Further surgery, following initial breast cancer surgery, is required in 25% - 30% of patients because of disease found at the edges of the tissue removed.

Reducing the need for further operations benefits patients (by reducing the number of operations required, improving cosmetic outcome and minimising anxiety) and the NHS (by realising economic benefits).

MarginProbe, a disposable probe which measures the margins of tissue removed during breast cancer surgery, allows the surgeon to remove further tissue during the same surgical procedure to clear any involved margins, minimising subsequent re-operations. Four hundred and sixty patients in 6 specialist Breast Units will be randomly allocated after BCS (and specimen radiology), by telephone randomisation, to either:

* MarginProbe assessment of the surgical specimen with re-excision of margins if required;
* Standard BCS (clinical and radiological clear margins) whereby the wound will be closed and the surgery completed (standard UK practice).

ELIGIBILITY:
Inclusion Criteria;

* Women aged 18-90 years with DCIS or Invasive Breast cancer containing DCIS diagnosed histopathologically.
* Histologically diagnosed DCIS or invasive lobular cancer in core biopsy (B5a or B5b).
* Tumour size 1.5cm - 4cm and undergoing breast cancer surgery. Written informed consent.

Exclusion Criteria;

* Unsuitable for BCS on basis of tumour size (<1.5cm or >4cm) or stage.
* Radiotherapy contraindicated.
* No histopathological evidence of DCIS or invasive lobular cancer.
* Neoadjuvant chemotherapy.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
To determine if intraoperative margin assessment after excision of a cancer reduces second operations (reexcision or mastectomy), compared to standard surgical practice by 9 months after primary surgery. | 9 months post surgery
  To determine if the use of the MarginProbe device, after surgical tumour excision and tissue specimen radiography of a breast cancer reduces rates of further surgical re-excision operations (re-excision or mastectomy), when compared to control/standard practice(whereby the wound is closed after radiography showing clear margins).

SECONDARY OUTCOMES:
Quality of Life | 9 months post surgery
  To determine the effect of checking for disease free tissue during the patients breast cancer surgery using the MarginProbe device (when compared to standard practice) on quality of life and Patient Related Outcome Measures.
EQ5D | 9 months post surgery
  To determine Quality of life and health related facility measures (EQ5D) between patient groups.
To compare the number of patients in both groups presenting with disease free margins greater than 1mm (circumferentially) after breast cancer surgery, using a laboratory histopathological assessment. | 9 months post surgery
  To compare the number of patients in both groups presenting with disease free margins greater than 1mm (circumferentially) after breast cancer surgery, using a laboratory histopathological assessment.
Total number of re-excisions | 9 months post surgery
  To compare the total number of re-excision procedures required in both groups (including mastectomy)following breast cancer surgery because of small (less than 1mm) disease free margins.
Cosmetic Outcome | 9 months post surgery
  Comparing digital photography assessment [2 views; front and side] to assess cosmetic outcomes in both study arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Peer Reviewed Scientific Journals Conference Presentation Publication on Website Access to raw data by Independent Steering Committee